CLINICAL TRIAL: NCT01329276
Title: A Randomized, Double-blind, Placebo-controlled, Two Way Cross-over Study to Assess the Particle Deposition and Acute Effects of Formoterol and Budesonide Combination Therapy (Symbicort® Forte Turbohaler®) on the Upper Airway Dimensions in COPD Patients.
Brief Title: Assess Particle Deposition and Acute Effects of Symbicort® Forte Turbohaler®) in COPD Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Wilfried A. De Backer, MD phD, University Hospital Antwerp
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PML_DOC_0905_/_ISSSYMB0020; 2009-016502-16 (EudraCT Number)
Record Dates: First submitted 2011-03-30; First posted 2011-04-05 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Symbicort; Turbohaler; Computational Fluid Dynamics; Functional Imaging; Budesonide; Formoterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Symbicort® forte Turbohaler® (Other)
  Interventions: Drug: Symbicort® forte Turbohaler®
- Placebo (lactose) (Placebo Comparator)
  Interventions: Drug: Symbicort® forte Turbohaler®

INTERVENTIONS:
Drug: Symbicort® forte Turbohaler® — 320 µg budesonide / 9 µg formoterol fumarate dihydrate

SUMMARY:
Computational Fluid Dynamics (CFD) is a new functional imaging method. Since CFD is very sensitive to detect small changes, it might be worthwhile to study the acute effect of formoterol and budesonide combination therapy (Symbicort® forte Turbohaler®) on the upper airway dimensions in severe COPD patients (GOLD III). The increased sensitivity of this technique makes it possible to detect changes in airway caliber in early stages. The regional distribution of resistance and the change in this parameter will provide more insight into the mode of action of the product.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented COPD based on the following criteria:

   Smoking history of at least 10 pack-years and decreased Tiffeneau index (FEV1/(F)VC < 0.70).
2. Patients should present severe COPD with an FEV1 between 50 and 30% of predicted (GOLD 3).
3. Male or female patients aged ≥ 40 years.
4. Patients should be treated according to GOLD guidelines before study start.
5. Patients with, in the opinion of the investigator, a co-operative attitude and ability to be trained to correctly use the TurbohalerR.
6. Maintained on stable respiratory medications for 6 weeks prior to visit 1.
7. Written informed consent obtained.

Exclusion Criteria:

1. Pregnancy, breast-feeding or planned pregnancy during the study. Fertile women not using acceptable contraceptive measures, as judged by the investigator.
2. Inability to carry out pulmonary function testing.
3. A respiratory infection or exacerbation of COPD in the four weeks prior to screening.
4. Any significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or influence the results of the study, or the patient's ability to participate in the study
5. A history of asthma, cystic fibrosis, central bronchiectasis, interstitial lung disease or pulmonary thromboembolic disease.
6. Cancer or any other chronic disease with poor prognosis and/or affecting patient status.
7. A history of thoracotomy with pulmonary resection.
8. Allergy, sensitivity or intolerance to study drugs and/or study drug formulation ingredients.
9. History of alcohol or drug abuse.
10. Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study.
11. Patients who received any investigational new drug within the last 4 weeks prior to the screening visit.
12. Patients treated with any non-permitted concomitant medication (see 7.2).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
total airway resistance
  To evaluate the effect of the combination therapy on the upper airway dimensions and to assess the particle deposition with Computational Fluid Dynamics (CFD). The parameters that will be obtained with CFD and used as primary outcome variables are total airway resistance and total airway volume.
total airway volume
  To evaluate the effect of the combination therapy on the upper airway dimensions and to assess the particle deposition with Computational Fluid Dynamics (CFD). The parameters that will be obtained with CFD and used as primary outcome variables are total airway resistance and total airway volume.

SECONDARY OUTCOMES:
effect of formoterol and budesonide combination therapy on lung function
  The secondary objective of this study is to assess the effect of formoterol and budesonide combination therapy on lung function (spirometry, body plethysmography and resistance).

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried A De Backer, MD PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem (Antwerp), Antwerp, Belgium